CLINICAL TRIAL: NCT00802126
Title: Efficacy of Combining Intravitreal Bevacizumab With Photodynamic Therapy Using Reduced Light Fluence Rate in Choroidal Neovascularization Secondary to Pathologic Myopia.
Brief Title: Intravitreal Bevacizumab and Low Fluence Photodynamic Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Chiosi Flavia, Chiosi Flavia, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81613
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and verteporfin (Experimental)
  Interventions: Drug: Combination therapy "IVB + rf-PDT"

INTERVENTIONS:
Drug: Combination therapy "IVB + rf-PDT" — low-fluence photodynamic therapy combined with intravitreal bevacizumab
  Other Names: Combined therapy: IVB + rf-PDT

SUMMARY:
The purpose of this study is to report the treatment effect and safety of combined intravitreal bevacizumab (IVB) and photodynamic therapy (PDT) with verteporfin using a reduced (RF) light fluence rate, in choroidal neovascularization (CNV) secondary to pathologic myopia.

DETAILED DESCRIPTION:
In this retrospective interventional case series, 16 patients with myopic CNV were included. All patients were treated with 1.25 mg of intravitreal bevacizumab followed by RF-PDT (25 J/cm²), 2 days later. All patients were previously treated with IVB monotherapy and active leaking of CNV occurred 90 to 120 days after the treatment.

Best-corrected visual acuity (BCVA-ETDRS), foveal thickness (FT) on optical coherence tomography (OCT), and fluorescein and indocyanine green angiographic (FA; ICG) findings were recorded. Follow-up evaluations were carried out for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Myopic CNV, CNV leakage

Exclusion Criteria:

* CNV not associated with high myopia
* No activity of CNV

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
BCVA improved | 6 months

SECONDARY OUTCOMES:
no CNV leakage | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Rinaldi, MD, PhD, Study Director — University of Campania Luigi Vanvitelli
Locations (1):
- Ophthalmology Department SUN, Napoli, Napoli, Italy